CLINICAL TRIAL: NCT00164190
Title: Trial of Routine Angioplasty and Stenting After Fibrinolysis to Enhance Reperfusion in Acute Myocardial Infarction- The TRANSFER-AMI Trial
Brief Title: Routine Angioplasty and Stenting After Fibrinolysis for Acute Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Heart Research Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Hoffmann-La Roche (Industry); Guidant Corporation (Industry)
Responsible Party: Dr. Warren Cantor, Canadian Heart Research Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCT-69798; FRN:69798
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2010-10-18 (Estimated); Status verified 2010-10

CONDITIONS: Myocardial Infarction
Keywords: Myocardial Infarction; Thrombolysis; Angioplasty; ST Elevation Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Routine Early Percutaneous Coronary Intervention after Thrombolysis — early or delayed PCI

SUMMARY:
Background:

In Canada, most patients with acute myocardial infarction (AMI) present to hospitals without cardiac catheterization facilities. Thrombolytic therapy remains the standard-of-care in these centres. However, thrombolytic therapy achieves normal coronary flow and myocardial perfusion in less than 50% of patients, and is associated with reocclusion, reinfarction, and recurrent ischemia. Primary angioplasty results in more complete reperfusion and lower rates of reocclusion, reinfarction and recurrent ischemia, but is not available in most centres. Although patients can be transferred for primary angioplasty, long transport times are associated with worse outcomes. An alternative strategy, described as facilitated angioplasty, involves administration of thrombolytic therapy at the community hospital followed by immediate transport for angioplasty. This approach achieves the benefits of primary angioplasty without delaying treatment. A well-conducted, prospective, randomized trial is needed to compare this strategy of facilitated angioplasty with standard thrombolytic therapy.

Objectives:

To evaluate the safety, feasibility, and efficacy of routine transfer of patients with AMI to an angioplasty centre immediately after thrombolysis for coronary angiography and percutaneous coronary intervention (PCI).

Hypothesis:

A strategy of routine transfer of patients with AMI to an angioplasty centre immediately after thrombolysis for coronary angiography and percutaneous intervention is associated with a significantly lower incidence of the composite of death, reinfarction, recurrent ischemia, heart failure, and shock at 30 days compared with the conventional strategy of thrombolysis with transfer reserved for failed reperfusion and/or development of shock.

Research Plan:

Patients with ST-elevation myocardial infarction and high-risk characteristics presenting to community hospitals without cardiac catheterization facilities will receive thrombolysis with tenecteplase and heparin (unfractionated or low molecular weight heparin) and will then be randomized to one of two strategies: facilitated PCI or standard treatment (thrombolysis with provisional rescue PCI). In the facilitated PCI group, patients will be transferred immediately to an angioplasty centre for urgent cardiac catheterization, and PCI if appropriate. In the standard treatment group, patients will only undergo urgent angiography for evidence of failed reperfusion and/or development of cardiogenic shock. The primary endpoint will be the composite of death, reinfarction, recurrent ischemia, heart failure, and shock at 30 days.

DETAILED DESCRIPTION:
Patients with ST-elevation myocardial infarction and high-risk characteristics presenting to community hospitals without cardiac catheterization facilities will receive thrombolysis with tenecteplase and heparin (unfractionated or low molecular weight heparin) and will then be randomized to one of two strategies: facilitated percutaneous coronary intervention (PCI) or standard treatment (thrombolysis with provisional rescue PCI). In the facilitated PCI group, patients will be transferred immediately to an angioplasty centre for urgent cardiac catheterization, and PCI if appropriate within 6 hours of thrombolysis. In the standard treatment group, patients will only undergo urgent angiography for evidence of failed reperfusion and/or development of cardiogenic shock.

ELIGIBILITY:
Inclusion Criteria:

1. Patients >= 18 years old who present within 12 hours of symptom onset with more than 30 minutes of continuous symptoms of an acute myocardial infarction to a centre that does not perform primary PCI, with either:

* >= 2 mm ST-segment elevation in 2 or more contiguous anterior leads
* >= 1 mm ST-segment elevation in 2 or more contiguous inferior leads with at least one of the following high-risk features:

  * Systolic blood pressure < 100 mm Hg
  * Heart rate > 100/minute
  * Killip Class II-III
  * >= 2 mm ST-segment depression in anterior leads
  * >= 1 mm ST-segment elevation in right-sided lead V4 (V4R), indicative of right ventricular involvement

Exclusion Criteria:

1. Left bundle branch block
2. Cardiogenic shock (Killip Class IV requiring vasopressors or inotropic support to maintain a systolic blood pressure > 90) prior to randomization
3. Active bleeding or known hemorrhagic diathesis
4. Availability of primary PCI with door-to-balloon time ≤ 60 minutes
5. Time from thrombolysis to initiation of consent process > 30 minutes
6. Use of thrombolytic agent other than tenecteplase (TNK) for index event
7. Major surgery, biopsy of parenchymal organ, or significant trauma in the past 6 weeks
8. Systolic blood pressure > 200 mm Hg or diastolic > 110 mm Hg after arrival to the hospital and before enrollment
9. Concomitant use of oral anticoagulants (e.g. warfarin) with International Normalized Ratio (INR) of > 2
10. Recent non-compressible vascular puncture
11. History of central nervous system structural damage (e.g. aneurysm, neoplasm, arteriovenous malformation, stroke) at any time, or transient ischemic attack within the last year
12. History of heparin-induced thrombocytopenia
13. Documented allergy to aspirin
14. Participation in other clinical research studies involving experimental therapies including drugs or devices within 7 days of enrollment or prior participation in this study
15. Inability to cooperate with the protocol or undergo cardiac catheterization
16. Other serious illness (e.g. active cancer, significant hepatic disease)
17. Serum creatinine > 140 umol/L
18. Percutaneous coronary intervention within one month
19. Previous bypass surgery
20. Pregnancy
21. Use of enoxaparin (or other low molecular weight heparin) in last 12 hours in patient > 75 years of age
22. Inferior ST-elevation myocardial infarction with none of the 5 high-risk features listed in the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2004-07; Primary Completion 2007-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
30-day composite of death (all cause) | 30 day
Reinfarction | 30 day
Recurrent ischemia | 30 day
New or worsening congestive heart failure, including readmission for heart failure | 30 day
Development of cardiogenic shock requiring inotropic support or intra-aortic balloon pump insertion | 30 day

SECONDARY OUTCOMES:
The incidence of major/severe bleeding, as defined by the thrombolysis in myocardial ischemia (TIMI) and Global Use of Strategies to Open Occluded Coronary Arteries (GUSTO) bleeding classifications in the first 30 days | 30 day
The proportion of patients with complete (> 70%) and partial (30-70%) ST-segment resolution from the qualifying electrocardiogram (ECG) to 6 hours after randomization | 30 day
Infarct size as assessed by QRS scoring system on the 180 minute 12-lead electrocardiogram | 30 day
The composite of death or reinfarction at 6 months | 30 day
The composite of death or reinfarction at 1 year | 30 day
Health costs | 30 day

CONTACTS AND LOCATIONS:
Overall Officials: Warren J. Cantor, MD, Principal Investigator — Caribbean Health Research Council
Locations (1):
- Southlake Regional Health Centre, Newmarket, Ontario, Canada

REFERENCES:
- [Derived] Arbel Y, Ko DT, Yan AT, Cantor WJ, Bagai A, Koh M, Eberg M, Tan M, Fitchett D, Borgundvaag B, Ducas J, Heffernan M, Morrison LJ, Langer A, Dzavik V, Mehta SR, Goodman SG; TRANSFER-AMI Trial Investigators. Long-term Follow-up of the Trial of Routine Angioplasty and Stenting After Fibrinolysis to Enhance Reperfusion in Acute Myocardial Infarction (TRANSFER-AMI). Can J Cardiol. 2018 Jun;34(6):736-743. doi: 10.1016/j.cjca.2018.02.005. Epub 2018 Feb 10. PMID 29801739
- [Derived] Russo JJ, Goodman SG, Cantor WJ, Tan MK, Borgundvaag B, Fitchett D, Dzavik V, Yan RT, Graham JJ, Mehta SR, Yan AT; TRANSFER-AMI Investigators. Efficacy and safety of a routine early invasive strategy in relation to time from symptom onset to fibrinolysis (a subgroup analysis of TRANSFER-AMI). Am J Cardiol. 2015 Apr 15;115(8):1005-12. doi: 10.1016/j.amjcard.2015.01.533. Epub 2015 Jan 31. PMID 25711435
- [Derived] Russo JJ, Goodman SG, Cantor WJ, Fitchett D, Heffernan M, Borgundvaag B, Ducas J, Cohen EA, Dzavik V, Mehta SR, Buller CE, Yan AT; TRANSFER-AMI investigators. Efficacy and safety of a routine early invasive strategy after fibrinolysis stratified by glycoprotein IIb/IIIa inhibitor use during percutaneous coronary intervention: a pre-specified subgroup analysis of the TRANSFER-AMI randomised controlled trial. Heart. 2014 Jun;100(11):873-80. doi: 10.1136/heartjnl-2013-305231. Epub 2014 Jan 21. PMID 24449716
- [Derived] Bagai A, Cantor WJ, Tan M, Tong W, Lamy A, Fitchett D, Cohen EA, Mehta SR, Borgundvaag B, Ducas J, Heffernan M, Dzavik V, Morrison L, Schwartz B, Lazzam C, Langer A, Goodman SG. Clinical outcomes and cost implications of routine early PCI after fibrinolysis: one-year follow-up of the Trial of Routine Angioplasty and Stenting after Fibrinolysis to Enhance Reperfusion in Acute Myocardial Infarction (TRANSFER-AMI) study. Am Heart J. 2013 Apr;165(4):630-637.e2. doi: 10.1016/j.ahj.2012.12.016. Epub 2013 Feb 19. PMID 23537982
- [Derived] Bhan V, Cantor WJ, Yan RT, Mehta SR, Morrison LJ, Heffernan M, Fitchett D, Dzavik V, Ducas J, Borgundvaag B, Cohen EA, Goodman SG, Yan AT. Efficacy of early invasive management post-fibrinolysis in men versus women with ST-elevation myocardial infarction: a subgroup analysis from Trial of Routine Angioplasty and Stenting after Fibrinolysis to Enhance Reperfusion in Acute Myocardial Infarction (TRANSFER-AMI). Am Heart J. 2012 Sep;164(3):343-50. doi: 10.1016/j.ahj.2012.05.022. Epub 2012 Aug 17. PMID 22980300
- [Derived] Lavi S, Cantor WJ, Casanova A, Tan MK, Yan AT, Dzavik V, Fitchett D, Cohen EA, Borgundvaag B, Heffernan M, Ducas J, Goodman SG. Efficacy and safety of enoxaparin compared with unfractionated heparin in the pharmacoinvasive management of acute ST-segment elevation myocardial infarction: Insights from the TRANSFER-AMI trial. Am Heart J. 2012 Feb;163(2):176-81.e2. doi: 10.1016/j.ahj.2011.10.015. PMID 22305834
- [Derived] Yan AT, Yan RT, Cantor WJ, Borgundvaag B, Cohen EA, Fitchett DH, Dzavik V, Ducas J, Tan M, Casanova A, Goodman SG; TRANSFER-AMI Investigators. Relationship between risk stratification at admission and treatment effects of early invasive management following fibrinolysis: insights from the Trial of Routine ANgioplasty and Stenting After Fibrinolysis to Enhance Reperfusion in Acute Myocardial Infarction (TRANSFER-AMI). Eur Heart J. 2011 Aug;32(16):1994-2002. doi: 10.1093/eurheartj/ehr008. Epub 2011 Feb 8. PMID 21307037
- [Derived] Cantor WJ, Fitchett D, Borgundvaag B, Ducas J, Heffernan M, Cohen EA, Morrison LJ, Langer A, Dzavik V, Mehta SR, Lazzam C, Schwartz B, Casanova A, Goodman SG; TRANSFER-AMI Trial Investigators. Routine early angioplasty after fibrinolysis for acute myocardial infarction. N Engl J Med. 2009 Jun 25;360(26):2705-18. doi: 10.1056/NEJMoa0808276. PMID 19553646